CLINICAL TRIAL: NCT01616966
Title: Laryngeal Injuries After Removal of the Tracheal Tube: A Comparison Between Anesthesia With Sevoflurane and Intravenous Anesthesia With Propofol A Randomized, Prospective, Controlled Trial
Brief Title: Laryngeal Injuries After Removal of the Tracheal Tube: A Comparison Between Sevoflurane and Propofol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rostock (Other)
Responsible Party: Principal Investigator, Thomas Mencke, Thomas Mencke, University of Rostock
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: A 2010 29
Record Dates: First submitted 2012-06-07; First posted 2012-06-12 (Estimated); Last update posted 2012-07-03 (Estimated); Status verified 2012-06

CONDITIONS: Vocal Cord; Injury, Superficial
Keywords: hoarseness; sore throat; vocal cord injuries
MeSH Terms: conditions — Wounds and Injuries; Hoarseness; Pharyngitis | interventions — Sevoflurane; Remifentanil; Propofol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sevoflurane (Active Comparator): Anesthesia was maintained with sevoflurane during surgery.
  Interventions: Drug: Sevoflurane
- Anesthesia with propofol (Active Comparator): Anesthesia was maintained with propofol during surgery.
  Interventions: Drug: propofol

INTERVENTIONS:
Drug: Sevoflurane — Maintenance of anesthesia with sevoflurane 1.0 Vol%
  Other Names: remifentanil
  Arms: Sevoflurane
Drug: propofol — Maintenance of anesthesia with propofol
  Other Names: remifentanil
  Arms: Anesthesia with propofol

SUMMARY:
Vocal cord injuries occur not only during tracheal intubation, but also during surgery and during removal of tracheal tube. Volatile anesthetics increase neuromuscular block of muscle relaxants. Thus, the investigators tested the hypothesis, that sevoflurane would cause less vocal cord injuries than a total intravenous anesthesia with propofol.

DETAILED DESCRIPTION:
Volatile anaesthetics increase neuromuscular block of neuromuscular blocking drugs. We tested the hypothesis, that sevoflurane would cause less vocal cord injuries than an intravenous anaesthesia with propofol. Sixty five patients were randomly assigned to the SEVO group (anaesthesia with sevoflurane) or TIVA group (anaesthesia with propofol). Vocal cord injuries were examined by stroboscopy before and 24 and 72 h after surgery; hoarseness was assessed up to 72 h.

ELIGIBILITY:
Inclusion Criteria:

* orotracheal intubation
* surgery of the ear
* written consent
* ASA I-III

Exclusion Criteria:

* preexisting pathologies of the vocal cords
* obesity
* difficult airway

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2010-08; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
incidence of vocal cord injuries | 24h after surgery
  assessed by stroboscopy

SECONDARY OUTCOMES:
incidence of hoarseness | 24h after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rostock, Rostock, Mecklenburg-Vorpommern, Germany